CLINICAL TRIAL: NCT05072327
Title: Mohs Surgery Combind With Cryotherapy for Eyelid Malignant Tumors: a Prospective Randomized Controlled Study.
Brief Title: Mohs Surgery Combind With Cryotherapy for Eyelid Malignant Tumors.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huasheng Yang, Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: yanghs20200921
Record Dates: First submitted 2021-10-03; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Eyelid Tumor
Keywords: Eyelid Tumor; Basal Cell Carcinoma; Squamous Cell Carcinoma; Sebaceous Carcinoma; Mohs surgery; cryotherapy
MeSH Terms: conditions — Eyelid Neoplasms; Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Adenocarcinoma, Sebaceous | interventions — Mohs Surgery; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mohs surgery conbind with cryotherapy (Experimental): patients in this group received both Mohs surgery and cryotherapy.
  Interventions: Procedure: Mohs surgery; Procedure: cryotherapy
- Mohs surgery (Active Comparator): patients in this group received only Mohs surgery.
  Interventions: Procedure: Mohs surgery

INTERVENTIONS:
Procedure: Mohs surgery — Mohs surgery of eyelid
Procedure: cryotherapy — cryotherapy of eyelid
  Arms: Mohs surgery conbind with cryotherapy

SUMMARY:
This study aim to investigate whether the prognosis of eyelid malignant tumor is better treated with Mohs surgery combind with cryotherapy than Mohs surgery only.

DETAILED DESCRIPTION:
This study is a randomized perspective study. American Joint Committee on Cancer was applied to define the cancer stage of patients recruited. Patients with Tis to T3cN0M0 will be randomized to receive Mohs surgery or Mohs suregery conbind cryotherapy. Patients will be followed for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of this study.
* Definite pathology signs of eyelid basal cell carcinoma, squamous cell carcinoma and sebacous carcinoma, Stage Tis to T3CN0M0 based on American Joint Committee on Cancer.
* Pathological examination showed the primary tumor was compeletely resected

Exclusion Criteria:

* Any previous treatment in the study eye
* Tumor complicated with infection
* Any other tumors of the paticipants
* Intolerate of surgery or anesthesia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
recurrence rate of tumor | three years
  measure the tumor recurrence rate for the two groups at three years
progression rate of tumor | three years
  measure the tumor progression rate for the two groups at three years

SECONDARY OUTCOMES:
all cause mortailty | three years
  measure the mortality rate for the two groups(Cancer-related death and non-Cancer-related death) at three years
side effects of Mohs surgery and cryotherapy in the treatment of eyelid malignant tumor | three years
  numbers of participants with side effects

CONTACTS AND LOCATIONS:
Overall Officials: Huasheng Yang, Doctor, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China